CLINICAL TRIAL: NCT04496375
Title: An Evaluation of Patients Access to Their Electronic Medical Records Via the IPC Connect Application
Acronym: ADN-CO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: ADN-CO-IPC 2020-004
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Solid Tumor; Hematologic Malignancy
Keywords: Electronic Medical Records; Patients anxiety
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Institut Paoli Calmettes Outpatients: Patients with a solid tumor or an hematologic malignancy who will attend an appointement at IPC Outpatients clinic
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Self-completed questionnaires

SUMMARY:
The aim of our study is to investigate the effect of providing patients access to their electronic medical records Via the IPC Connect Application on their A Survey will be proposed to all outpatients with a solid or hematologic malignancy who will attend an appointement at Institut Paoli Calmettes clinic.

Data will be collected during a 1-month period. The auto-questionnaire will be composed of 31 questions addressed to all patients, 17 questions will be specifically addressed to patients using IPC connect application and 7 questions will be addressed to patients who do not use the application.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, age> 18 Years
* Solid tumor or hematologic malignancy
* Patient attending an appointment at Institut Paoli Calmettes
* Non-opposition

Exclusion Criteria:

* emergency, Vulnerable person or unable to provide informed consent
* First appointment at Institut Paoli Calmettes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All outpatients with an solid tumor or an hematologic malignancy who will attend Institut Paoli-Calmettes Outpatients clinic during 1 months
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2020-11-05 (Estimated); Primary Completion 2020-12-05 (Estimated); Study Completion 2020-12-05 (Estimated)

PRIMARY OUTCOMES:
Impact of Patients Access to Their Electronic Medical Records Via the IPC Connect Application on patients anxiety level | 1 day
  Anxiety level will be measured by the Hospital Anxiety and Depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle Gravis, Principal Investigator — Institut Paoli-Calmettes

IPD SHARING:
Plan to Share IPD: No